CLINICAL TRIAL: NCT00374686
Title: Prophylactic Vs Preemptive Oral Valganciclovir for Management of Cytomegalovirus Infection in Adult Renal Transplant Recipients: A Clinical and Pharmacoeconomic Study
Brief Title: Study of Prophylactic Vs Preemptive Valganciclovir
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Hoffmann-La Roche (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VAL015 HSC02-0140
Record Dates: First submitted 2006-09-07; First posted 2006-09-11 (Estimated); Last update posted 2006-09-11 (Estimated); Status verified 2005-09

CONDITIONS: Cytomegalovirus Infection
Keywords: cytomegalovirus; kidney; transplantation; valganciclovir; preemptive
MeSH Terms: conditions — Cytomegalovirus Infections | interventions — Valganciclovir

INTERVENTIONS:
Drug: Valganciclovir

SUMMARY:
This is a study of prophylactic Vs preemptive oral valganciclovir for management of cytomegalovirus infection in adult renal transplant recipients looking at clinical and pharmacoeconomic outcomes

DETAILED DESCRIPTION:
This is a study of prophylactic Vs preemptive oral valganciclovir for management of cytomegalovirus infection in adult renal transplant recipients looking at clinical and pharmacoeconomic outcomes. Patients at risk for CMV (D+/R-, D+/R+, D-/R+) were randomized to prophylaxis (valganciclovir 900 mg qd for 100 days, n=49) or preemptive therapy (900 mg bid for 21 days, n=49) for CMV DNAemia (CMV DNA level >2000 copies/ml in ≥ 1 whole blood specimens by quantitative PCR done weekly for 16 weeks then at months 5, 6, 9, and 12. Clinical and virologic outcomes were measured and pharmacoeconomic outcomes will be analyzed

ELIGIBILITY:
Inclusion Criteria:

* All patients who received a kidney transplant at Washington University Medical Center between March 2003 and June 2004.

Exclusion Criteria:

* Age younger than 18
* Refusal to consent for the study
* Allergy to ganciclovir and severe illness too serious to justify randomization

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2003-03; Study Completion 2005-09

PRIMARY OUTCOMES:
Primary outcomes included occurrence of CMV infection and disease and response to therapy

SECONDARY OUTCOMES:
Secondary outcomes were incidence of acute rejection, allograft survival, allograft dysfunction, death, and incidence of neutropenia

CONTACTS AND LOCATIONS:
Overall Officials: Daniel C Brennan, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Result] Khoury JA, Storch GA, Bohl DL, Schuessler RM, Torrence SM, Lockwood M, Gaudreault-Keener M, Koch MJ, Miller BW, Hardinger KL, Schnitzler MA, Brennan DC. Prophylactic versus preemptive oral valganciclovir for the management of cytomegalovirus infection in adult renal transplant recipients. Am J Transplant. 2006 Sep;6(9):2134-43. doi: 10.1111/j.1600-6143.2006.01413.x. Epub 2006 Jun 19. PMID 16780548
- [Derived] Vernooij RW, Michael M, Colombijn JM, Owers DS, Webster AC, Strippoli GF, Hodson EM. Pre-emptive treatment for cytomegalovirus viraemia to prevent cytomegalovirus disease in solid organ transplant recipients. Cochrane Database Syst Rev. 2025 Jan 14;1(1):CD005133. doi: 10.1002/14651858.CD005133.pub4. PMID 39807668
- [Derived] Vernooij RW, Michael M, Ladhani M, Webster AC, Strippoli GF, Craig JC, Hodson EM. Antiviral medications for preventing cytomegalovirus disease in solid organ transplant recipients. Cochrane Database Syst Rev. 2024 May 3;5(5):CD003774. doi: 10.1002/14651858.CD003774.pub5. PMID 38700045